CLINICAL TRIAL: NCT04778124
Title: Safety and Effectiveness of Hemorrhoidal Artery Ligation Using the HAL-RAR Technique for Hemorrhoidal Disease
Brief Title: HAL-RAR Technique for Treating Hemorrhoids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amalia Fleming General Hospital (Other)
Collaborators: Sismanoglio - Amalia Fleming General Hospital (Unknown)
Responsible Party: Principal Investigator, Georgia Dedemadi, MD, PhD, FACS, Amalia Fleming General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2042/4-3-2020
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Hemorrhoidal Disease
Keywords: hemorrhoidal disease; treatment; HAL; RAR; mucopexy
MeSH Terms: interventions — Hemorrhoidectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with hemorrhoidal disease undergoing HAL-RAR (Other): This is a single-arm trial, in which all patients with grade II hemorrhoidal disease resistant to conservative treatment, grade III and IV hemorrhoidal disease underwent HAL RAR surgery.
  Interventions: Procedure: Hemorrhoidal Arterial Ligation (HAL) and Recto Anal Repair (RAR); Procedure: Excision of thrombosed hemorrhoid / Hemorrhoidectomy /

INTERVENTIONS:
Procedure: Hemorrhoidal Arterial Ligation (HAL) and Recto Anal Repair (RAR) — All patients underwent hemorrhoidal artery ligation on multiple sites according to pulsations detected by the doppler transducer and mucopexy (RAR) at the sites of prolapse.
Procedure: Excision of thrombosed hemorrhoid / Hemorrhoidectomy / — One patient with mucosal necrosis of the hemorrhoidal cushion postoperatively underwent hemorrhoidectomy with excision of necrotic tissues.Furthermore, 2 patients who presented with hemorrhoidal thrombosis postoperatively underwent emergency surgery with supplementary excision of the thrombosed hemorrhoid. In addition, 9 patients who experienced recurrence of hemorrhoidal disease after undergoing HAL-RAR surgery, were treated with hemorrhoidectomy according to the Milligan-Morgan procedure.

SUMMARY:
A wide variety of methods has been proposed for treating hemorrhoidal disease with excisional hemorrhoidectomy remaining the gold standard. The aim of this trial is to assess the safety and effectiveness of the HAL-RAR technique in treating hemorrhoidal disease. Arterial ligation was performed by using the highest doppler signal to locate the site of the hemorrhoidal artery in combination with RAR in order to reposition redundant rectal mucosa/submucosa that prolapses to its original anatomical location, leading to resolution of symptoms.

This is a retrospective study from January 2010 to November 2019 of patients who underwent HAL-RAR for hemorrhoidal disease. Demographics, degree of disease, length of hospital stay, postoperative pain, complications (urinary retention, dyschezia, bleeding, necrosis of a hemorrhoid, anal discomfort, sensation of fullness) and recurrence were recorded. Patients were followed-up at postoperative day 1 and 8, and at 1, 6 and 12 months. The main outcome of the study was recurrence. Secondary outcomes included postoperative complications, postoperative pain and patient-assessed resolution of symptoms.

DETAILED DESCRIPTION:
This is a retrospective, single-institution, study conducted from January 2010 to November 2019. Grade of hemorrhoidal disease was assessed according to Goligher's classification. Patients with grade II, resistant to conservative treatment, grade III and IV hemorrhoidal disease that underwent the HAL-RAR technique, were included in the study. Patients with grade II disease presented a small degree of prolapse. Non-surgical techniques, such as rubber-band ligation or injection of sclerosing agents, were not performed prior to the HAL-RAR operation since this is not a common practice in our institution. Conservative treatment for grade II hemorrhoids included diet rich in fiber, lifestyle modifications (increased fluid intake, improved anal hygiene, avoiding staining and constipation), the use of phlebotonics and other topical ointments that contained a combination of local anesthetics, corticosteroids and antiseptics, designed to relieve symptoms of pruritus and discomfort.

The study was reviewed and approved by the institution's ethics committee. Detailed informed consent was obtained from all patients before the operative procedure. Exclusion criterion included age <18 years, pregnancy, coagulation disorders, patients with major comorbidities (American Society of Anesthesiologists [ASA] ≥3), psychiatric conditions preventing collaboration and follow-up, other concomitant anorectal disease (rectal prolapse, anal fissure, anal stenosis, perianal fistula or abscess, fecal incontinence) and previous pelvic radiotherapy. Preoperative clinical assessment and classification for all patients included complete medical history particularly underlining hemorrhoidal disease-related symptoms, physical examination, proctoscopy, and rigid sigmoidoscopy. Further investigation was performed when necessary.

Demographic data, degree of hemorrhoidal disease, length of hospital stay, perioperative and postoperative data were recorded. Clinical assessment and surgery were performed by two of the authors trained and experienced with the technique. Patients did not receive a solid diet after 10:00p.m. the night before surgery. Preoperative preparation included one or two phosphate enemas before the procedure. Antibiotic prophylaxis was not considered mandatory and was not administered. The severity of pain was self-evaluated by the patients using a visual analogue scale (VAS) with 0 indicating the absence of pain and 10 the worst possible pain. Data about analgesic consumption was also recorded. Postoperatively, intravenous Paracetamol 3gr and Parecoxid 80mg was administered daily, and in cases of severe pain Tramadol 500mg was given upon request. Patients were discharged when adequate pain control was achieved. They were examined by the surgeon to rule out early complications and ensure the outcome of the operation. Patients were advised to avoid prolonged straining and heavy physical activity for 1 month and to consume at least 2 liters of water per day and a diet rich in fiber, supplemented by the oral consumption of stool softeners. After discharge, oral analgesics were prescribed that consisted of nonsteroidal anti-inflammatory agents and oral narcotics. Patients were followed-up on postoperative day 1 and 8, and at 1, 6 and 12 months and evaluated with a proctologic examination. A patient directed diary card to assess the resolution of symptoms was implemented. Recurrence was evaluated after physical examination and defined as relapse of symptoms such as bleeding or prolapse often daily requiring manual reduction. The main outcome of the study was recurrence. Secondary outcomes included postoperative complications, postoperative pain and patient-assessed resolution of symptoms. Continuous variables are presented as median values and range, and categorical variables, as numbers and percentages.

Surgical technique The operation was performed, with the patient in the lithotomy position, under general or spinal anesthesia according to the patient's preference in consultation with the anesthesiologist. Perianal block was not offered as an alternative. The region is then treated with an antiseptic solution. After lubrication with xylocaine gel, the anal canal is dilated to a width of two fingers to allow insertion of the proctoscope. The HAL proctoscope, equipped with a doppler transducer (HAL II Doppler, A.M.I., Feldkirch, Austria) which is orientated just below the proctoscope's lateral ligation window, allows the identification and the selective ligation of the hemorrhoidal artery. In addition, a built-in light source provides illumination for easy placement of sutures under direct vision. As the submucosal terminal branches of the superior hemorrhoidal artery are best identified with the Doppler signal 2cm above the dentate line, the proctoscope was inserted 5-6 cm above the anal verge for best localization. The operation started and ended at the 12 o'clock position. The proctoscope was then rotated clockwise in search of the 6 main terminal branches, usually located at 1, 3, 5, 7, 9 and 11 o'clock. Once identified, the proctoscope was slowly withdrawn distally until the best Doppler signal was obtained. Arterial ligation was then performed with a "Z" suture using 2-0 polyglycolic acid and 5/8-inch needle. A knot-pusher was used to secure the suture. The lateral ligation window in the proctoscope's lumen was used to calculate the exact depth of the transfixed sutures. By inserting the tip of the needle holder inside the pivot hole before suturing, it ensured a maximum depth of 6mm, primarily involving the mucosa and submucosa, avoiding the perforation of the entire rectal wall. Eradication or significant reduction of the Doppler signal when tying the suture confirmed the successful arterial ligation. The proctoscope was rotated clockwise at the same level to locate further arteries. Once a full rotation had been completed, the procedure was repeated 15mm below the first series of sutures. The number of arterial ligations ranged from 6 to 10. After completion of the arterial ligation the RAR procedure, known as mucopexy, was performed where hemorrhoidal prolapse was detected. Using the same proctoscope, the outer sleeve is removed, in order to expand the operating window and expose a wider rectal mucosal area. The prolapsing tissue comes under direct vision inside the proctoscope's lumen. RAR is carried out with a continuous suture along the longitudinal axis in a proximal-to-distal direction in the lower part of the rectum with the same 2-0 polyglycolic acid and 5/8-inch needle. The continuous suture of the mucosa and submucosa can be performed repeatedly according to the size and extent of the prolapse and must always entrap the site of the hemorrhoidal artery with suture above and below. It is important to ensure 5mm distance between each suture, to avoid tissue ischemia and ensure sufficient venous outflow from the hemorrhoids. The continuous suture ends up to 1cm proximal to the dentate line, sparing the anal canal, avoiding postoperative pain. After securing the continuous suture the redundant rectal mucosa/submucosa that prolapses is repositioned to its original anatomical location. The number of RAR performed ranged from 1 to 5, while special attention was given to stay above the dentate line.

ELIGIBILITY:
Inclusion Criteria:

Patients with

* grade II hemorrhoidal disease, resistant to conservative treatment
* grade III hemorrhoidal disease,
* grade IV hemorhoidal disease,

that underwent the HAL-RAR technique.

Exclusion Criteria:

* pregnancy
* coagulation disorders
* patients with major comorbidities (American Society of Anesthesiologists [ASA] ≥3),
* psychiatric conditions preventing collaboration and follow-up
* other concomitant anorectal disease (rectal prolapse, anal fissure, anal stenosis, perianal fistula or abscess, fecal incontinence)
* previous pelvic radiotherapy
* declined consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Recurrence | Postoperatively at 1 month
  Recurrence was evaluated after physical examination and defined as a relapse of symptoms such as bleeding or prolapse often daily requiring manual reduction.
Recurrence | Postoperatively at 6 months
  Recurrence was evaluated after physical examination and defined as a relapse of symptoms such as bleeding or prolapse often daily requiring manual reduction.
Recurrence | Postoperatively at 12 months
  Recurrence was evaluated after physical examination and defined as a relapse of symptoms such as bleeding or prolapse often daily requiring manual reduction.

SECONDARY OUTCOMES:
Postoperative complications | Postoperative day 1
  Postoperative compications included urinary retention,dyschezia,bleeding, necrosis of a hemorrhoid,remnant symptoms such as anal discomfort and sensation of fullness
Postoperative complications | Postoperative day 8
  Postoperative compications included urinary retention,dyschezia,bleeding, necrosis of a hemorrhoid,remnant symptoms such as anal discomfort and sensation of fullness
Postoperative complications | Postoperatively at 1 month
  Postoperative compications included urinary retention,dyschezia,bleeding, necrosis of a hemorrhoid,remnant symptoms such as anal discomfort and sensation of fullness
Postoperative pain | Postoperative day 1
  Pain was self-evaluated by the patients using a visual analogue scale (VAS) with 0 indicating the absence of pain and 10 the worst possible pain.
Postoperative pain | Postoperative day 8
  Pain was self-evaluated by the patients using a visual analogue scale (VAS) with 0 indicating the absence of pain and 10 the worst possible pain.
Postoperative pain | Postoperatively at 1 month
  Pain was self-evaluated by the patients using a visual analogue scale (VAS) with 0 indicating the absence of pain and 10 the worst possible pain.
Patient-assessed resolution of symptoms | Postoperative day 1
  A patient directed diary card to assess the resolution of symptoms was implemented.
Patient-assessed resolution of symptoms | Postoperative day 8
  A patient directed diary card to assess the resolution of symptoms was implemented.
Patient-assessed resolution of symptoms | Postoperatively at 1 month
  A patient directed diary card to assess the resolution of symptoms was implemented.
Patient-assessed resolution of symptoms | Postoperatively at 6 months
  A patient directed diary card to assess the resolution of symptoms was implemented.
Patient-assessed resolution of symptoms | Postoperatively at 12 months
  A patient directed diary card to assess the resolution of symptoms was implemented.

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Dedemadi, MD, PhD, Principal Investigator — Amalia Fleming Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morinaga K, Hasuda K, Ikeda T. A novel therapy for internal hemorrhoids: ligation of the hemorrhoidal artery with a newly devised instrument (Moricorn) in conjunction with a Doppler flowmeter. Am J Gastroenterol. 1995 Apr;90(4):610-3. PMID 7717320
- [Background] Ratto C, Campenni P, Papeo F, Donisi L, Litta F, Parello A. Transanal hemorrhoidal dearterialization (THD) for hemorrhoidal disease: a single-center study on 1000 consecutive cases and a review of the literature. Tech Coloproctol. 2017 Dec;21(12):953-962. doi: 10.1007/s10151-017-1726-5. Epub 2017 Nov 24. PMID 29170839
- [Background] Popov V, Yonkov A, Arabadzhieva E, Zhivkov E, Bonev S, Bulanov D, Tasev V, Korukov G, Simonova L, Kandilarov N, Taseva A, Dimitrova V. Doppler-guided transanal hemorrhoidal dearterilization versus conventional hemorrhoidectomy for treatment of hemorrhoids - early and long-term postoperative results. BMC Surg. 2019 Jan 10;19(1):4. doi: 10.1186/s12893-019-0469-9. PMID 30630463
- [Background] Aigner F, Gruber H, Conrad F, Eder J, Wedel T, Zelger B, Engelhardt V, Lametschwandtner A, Wienert V, Bohler U, Margreiter R, Fritsch H. Revised morphology and hemodynamics of the anorectal vascular plexus: impact on the course of hemorrhoidal disease. Int J Colorectal Dis. 2009 Jan;24(1):105-13. doi: 10.1007/s00384-008-0572-3. Epub 2008 Sep 3. PMID 18766355
- [Background] Gallo G, Martellucci J, Sturiale A, Clerico G, Milito G, Marino F, Cocorullo G, Giordano P, Mistrangelo M, Trompetto M. Consensus statement of the Italian society of colorectal surgery (SICCR): management and treatment of hemorrhoidal disease. Tech Coloproctol. 2020 Feb;24(2):145-164. doi: 10.1007/s10151-020-02149-1. Epub 2020 Jan 28. PMID 31993837
- [Background] Emile SH, Elfeki H, Sakr A, Shalaby M. Transanal hemorrhoidal dearterialization (THD) versus stapled hemorrhoidopexy (SH) in treatment of internal hemorrhoids: a systematic review and meta-analysis of randomized clinical trials. Int J Colorectal Dis. 2019 Jan;34(1):1-11. doi: 10.1007/s00384-018-3187-3. Epub 2018 Nov 12. PMID 30421308
- [Derived] Karkalemis K, Chalkias PL, Kasouli A, Chatzaki E, Papanikolaou S, Dedemadi G. Safety and effectiveness of hemorrhoidal artery ligation using the HAL-RAR technique for hemorrhoidal disease. Langenbecks Arch Surg. 2021 Nov;406(7):2489-2495. doi: 10.1007/s00423-021-02190-0. Epub 2021 May 6. PMID 33959805